CLINICAL TRIAL: NCT01197183
Title: Survey for the Initial Treatment of Hypothyroidism in France
Brief Title: Observational Study With Prospective and/or Retrospective Follow-up, Without Modifying Patient Treatment and Follow-up Practices for the Initial Treatment of Hypothyroidism in France
Acronym: ORCHIDEE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr. Frederic Landron, Laboratoires Merck Lipha Santé, an affiliate of Merck KGaA, Darmstadt, Germany
Other Study IDs: 200007-502
Record Dates: First submitted 2010-08-18; First posted 2010-09-09 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2010-09

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Thyroid hormones
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

SUMMARY:
This observational survey with prospective and/or retrospective follow-up is designed to study practices for the initial treatment of hypothyroidism in France without modifying subject treatment.

DETAILED DESCRIPTION:
Thyroid disorder can be central, caused by a deficiency in thyroid stimulating hormone (TSH) production; or peripheral, caused by the decrease in the plasma concentration of thyroid hormones, more specifically of free thyroxine (free T4). Peripheral hypothyroidism is caused by the decrease in the production capacities of the thyroid gland.

The treatment of hypothyroidism is based on the restoration and maintenance of biological (judged on the basis of the standardised TSH and T4 values) and clinical euthyroidism.

A number of forms of thyroid hormones are available in the French market (Euthyral®, Cynomel®, L-thyroxine drops®), of which, Levothyrox® is the most frequently prescribed drug in this category.

The treatment of peripheral hypothyroidism, in particular, is well codified and almost consensual. In France, there is no published observational study, based on which one can document the manner in which subjects are treated. This observational study is set up to document these practices.

OBJECTIVES The principal objectives of this survey is to to get information on the use of Levothyrox in France

* Circumstances of diagnosis
* Record realised
* Terms and conditions of treatment by the general practitioner and/or the endocrinologist

The secondary objective is to evaluate the inclusion criteria for levothyroxine treatment.

For each subject the participating doctor will complete a follow up questionnaire form until the first control level of TSH after the diagnosis of hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed hypothyroid subject (either during the inclusion period, or within the 6 previous months) for whom, data related to the diagnosis is available if the diagnosis was not carried out initially by the investigating doctor
* Subject, who has given his/her oral consent for participation

Exclusion Criteria:

* Subject included in clinical trial or having participated in a clinical trial during the last 3 months
* Subject presenting a major and objectifiable risk of not being able to follow-up until the next TSH level (moving, problems encountered during another study, pathology affecting the vital prognosis in the short-term)
* All contraindications to Lévothyrox

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Independent, hospital and mixed practice endocrinologists and general practitioners enrolled 1000 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1285 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Initial questionnaire | Baseline
  Documentation of indications for levothyroxine treatment

SECONDARY OUTCOMES:
Follow-up questionnaire | 3 months
  Documentaion of inclusion criteria (socio-demographic and clinical data, treatment information and biological values) for levothyroxine treatment. Follow-up questionnaire filled-in until the result of the first TSH level after commencement of therapy with thyroid hormones.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Frederic Landron, MD, Study Director — Laboratoires Merck Lipha Santé
Locations (1):
- Merck Lipha Santé Laboratories, Saint-Romain, Lyon, France